CLINICAL TRIAL: NCT04508881
Title: To Compare the Intraluminal Stenting and External Ligation of Ahmed Glaucoma Valve (AGV) Regarding Refractory Glaucoma Management and Postoperative Hypotony Prevention.
Brief Title: Intraluminal Stenting Versus External Ligation of Ahmed Glaucoma Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Faried Mohammed Wagdy, Doctor of Ophthalmolgy- Menoufia hospital, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Faried1976; Tharwat Mokbel (Other: Mansoura univerity)
Record Dates: First submitted 2020-07-21; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: : This randomized clinical trial included 30 eyes of 25 patients (age range: 44-56 y) with refractory glaucoma. This study was conducted during the period from September 2018 to January 2020. The study included two groups, AGV with intraluminal stenting group (n=15) and AGV with external ligation group (n=15). Follow up continued to a year post operation. The primary outcome was Intraocular pressure (IOP) and its association with the number of postoperative glaucoma medications. IOP ≤ 21 mmHg without medications announced complete success while IOP ≤ 21 mmHg with medications indicated qualified success. IOP of <6 mmHg defined hypotony.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External ligation (Active Comparator): External ligation of the valve tube by vicryl sutures
  Interventions: Device: Ahmed Glaucoma Valve
- intraluminal stenting (Active Comparator): stenting of the valve tube by prolene suture
  Interventions: Device: Ahmed Glaucoma Valve

INTERVENTIONS:
Device: Ahmed Glaucoma Valve — To compare the prevalence of postoperative hypotony between the 2 arms

SUMMARY:
Objectives: To compare the intraluminal stenting and external ligation of Ahmed Glaucoma Valve (AGV) regarding refractory glaucoma management and postoperative hypotony prevention.

Patients and Methods: This randomized clinical trial included 30 eyes of 25 patients (age range: 44-56 y) with refractory glaucoma. This study was conducted during the period from September 2018 to January 2020. The study included two groups, AGV with intraluminal stenting group (n=15) and AGV with external ligation group (n=15). Follow up continued to a year post operation. The primary outcome was Intraocular pressure (IOP) and its association with the number of postoperative glaucoma medications. IOP ≤ 21 mmHg without medications announced complete success while IOP ≤ 21 mmHg with medications indicated qualified success. IOP of <6 mmHg defined hypotony.

Key Words: Stenting- ligation- Ahmed valve- Hypotony

DETAILED DESCRIPTION:
Introduction: Refractory glaucoma is a complicated type of glaucoma difficult to be treated. This type is characterized by high IOP with a high resistance to be reduced by traditional medical or surgical therapy. Shunt surgery improve trabeculectomy poor long term outcomes in refractory glaucoma.1 AGV, a shunt device, is used either from the start or after conventional procedures failure in refractory glaucoma. It helps the aqueous humour flow direct in the silicone tube.2 AGV is effective in reducing the postoperative hypotony commonly seen in non valved implants however the presence of persistent hypotony is still a problem after AGV.3 Persistent hypotony after AGV is caused by over-priming the tube and excessive manipulation of the valve housing that may damage the valve mechanism, the outflow of aqueous humour around the silicone tube immediately post-operatorive after the utilization of a 22 or 23G needle in creation of the sclerostomy and ciliary body function failure post-surgery in complicated eyes in which AGV is used. 4-5 closure of the tube by ligation or stenting may be needed when postoperative ocular hypotony occurs. 6 Enough and expected outflow control may not be induced by ligation of the tube at a focal area. 7 postoperative ocular hypotony could be managed effectively by Ab interno tube stenting. 8-10 Patients and Methods: Thirty eyes with refractory glaucoma were included in randomized controlled clinical trial. Patients aged from 44 to 56 years old. Despite of tolerated medication after previous trabeculectomy surgery, those patients had high intraocular pressure (IOP). Approval of institutional research board committee was taken. Two groups were studied; AGV with intraluminal stenting group (n=15 eyes) and AGV with external ligation group (n=15 eyes). Follow- up to one year after the surgery was done. The primary outcome was Intraocular pressure (IOP) and its association with the number of postoperative glaucoma medications. IOP ≤ 21 mmHg without medications announced complete success while IOP ≤ 21 mmHg with medications indicated qualified success. IOP of <6 mmHg defined hypotony. All patients preoperatively were subjected to IOP measurement using Goldman applanation tonometer, visual acuity assessment (VA) using Snellen E chart, visual field analysis (VF) by Humphrey visual field analyzer, Angle examination by goniolens, optic disc examination by Volk+90 lens, sit lamp examination for assessment of corneal clarity and any corneal touch with the tube and anterior chamber depth. All patients had peribulbar anaesthesia. Operative technique: in group I, incision of superior-temporal conjunctiva was carried out, appropriate cauterization and approximately at 10 mm posterior to the corneal limbus, the valve body plate was placed. Forceps was used to insert A 7-0 prolene thread into the tube lumen; the prolene 7-0 thread was cut with scissors making it along the tube length to remove it when needed. (Figure 2) In group II, the same as in group I but 8-0 vicryl was used to ligate the tube with the underlying sclera in addition to usage of two interrupted prolene 7-0 sutures applied 2mm apart over the tube itself to make partial occlusion and then entered into the anterior chamber. (Figure 3) Postoperative treatment with combined antibiotic and steroid eye drops every four hours in the first week followed by 2 weeks gradual tapering. IOP, VA, VF, optic disc examination by Volk+90 lens, slit lamp examination were the follow-up parameters. Failure was considered if the patient needed to implant removal, added glaucoma surgery, or developed phthisis bulbi.

Statistical analysis: Data were statistically analyzed by SPSS version 22(SPSS Inc., Chicago, IL, USA). Non-paired t test and Mann-Whitney were applied to quantitative variables. Fisher's exact test was applied to qualitative variables. Correlation was used to assess strength and direction of association. Less than 0.05 P value was set to be significant.

Data Availability Statement:The data used to support the findings of this study are included within the article.

Compliance with Ethical Standards Funding Statement: None Conflicts of Interest: The author declares that there he has no conflict of interest regarding the publication of this paper.

Ethical approval: All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

Informed consent: Informed consent was obtained from all individual participants included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 30 eyes of 25 patients (age range: 44-56 y) with refractory glaucoma

Exclusion Criteria:

* other types of glaucoma

Ages: 44 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 1 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Postoperative hypotony | 1 year
  by measuring intraocular poressure postoperatively by Goldmann Applanation tonometer

SECONDARY OUTCOMES:
postoperative hypertensive phase by Goldmann Applanation tonometer | 1 year
  by studying the incidence of hypertensive phase postoperatively
low Complications | 1 year
  by slit lamp examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faried Wagdy, Cairo, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No